CLINICAL TRIAL: NCT06578832
Title: Assessment of The Oral Health Status of Children With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2022.961
Record Dates: First submitted 2024-08-25; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Caries,Dental; Quality of Life; Saliva Altered; Periodontitis
Keywords: Chronic kidney disease; oral health; salivary; quality of life
MeSH Terms: conditions — Renal Insufficiency, Chronic; Dental Caries; Periodontitis | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Children with chronic kidney disease: It is a group of patients between the ages of 4 and 17 who have recently been diagnosed with jchronic kidney disease
  Interventions: Diagnostic Test: physical and chemical methods; Diagnostic Test: biochemical methods; Diagnostic Test: biochemical tests; Diagnostic Test: Oral Health Habits; Diagnostic Test: Oral Findings; Diagnostic Test: Quality of Life Assessment
- Healthy patient group: Healthy children aged between 4 and 17 years, with no systemic diseases and not taking any regular medications.
  Interventions: Diagnostic Test: physical and chemical methods; Diagnostic Test: biochemical methods; Diagnostic Test: biochemical tests; Diagnostic Test: Oral Health Habits; Diagnostic Test: Oral Findings; Diagnostic Test: Quality of Life Assessment
- Children with chronic kidney disease receiving dialysis treatment: It is a group of patients aged between 4 and 17 who have recently been diagnosed with chronic kidney disease and are receiving dialysis treatment.
  Interventions: Diagnostic Test: physical and chemical methods; Diagnostic Test: biochemical methods; Diagnostic Test: biochemical tests; Diagnostic Test: Oral Health Habits; Diagnostic Test: Oral Findings; Diagnostic Test: Quality of Life Assessment
- Children with chronic kidney disease who have undergone a kidney transplant: It is a group of patients aged between 4 and 17 who have recently been diagnosed with chronic kidney disease and have undergone a kidney transplant.
  Interventions: Diagnostic Test: Oral Health Habits; Diagnostic Test: Oral Findings; Diagnostic Test: Quality of Life Assessment
- Children with stage 1-3 chronic kidney disease: It is a group of patients aged between 4 and 17 who have been diagnosed with stage 1-3 chronic kidney disease
  Interventions: Diagnostic Test: physical and chemical methods; Diagnostic Test: biochemical methods; Diagnostic Test: biochemical tests; Diagnostic Test: Oral Health Habits; Diagnostic Test: Oral Findings; Diagnostic Test: Quality of Life Assessment
- Children with stage 4-5 chronic kidney disease: It is a group of patients aged between 4 and 17 who have been diagnosed with stage 4-5 chronic kidney disease
  Interventions: Diagnostic Test: physical and chemical methods; Diagnostic Test: biochemical methods; Diagnostic Test: biochemical tests; Diagnostic Test: Oral Health Habits; Diagnostic Test: Oral Findings; Diagnostic Test: Quality of Life Assessment

INTERVENTIONS:
Diagnostic Test: physical and chemical methods — Salivary flow rate, pH, buffering capacity
  Groups: Children with chronic kidney disease; Children with chronic kidney disease receiving dialysis treatment; Children with stage 1-3 chronic kidney disease; Children with stage 4-5 chronic kidney disease; Healthy patient group
Diagnostic Test: biochemical methods — Total oxidant and antioxidant capacities
  Groups: Children with chronic kidney disease; Children with chronic kidney disease receiving dialysis treatment; Children with stage 1-3 chronic kidney disease; Children with stage 4-5 chronic kidney disease; Healthy patient group
Diagnostic Test: biochemical tests — urea, calcium, potassium, phosphorus
  Groups: Children with chronic kidney disease; Children with chronic kidney disease receiving dialysis treatment; Children with stage 1-3 chronic kidney disease; Children with stage 4-5 chronic kidney disease; Healthy patient group
Diagnostic Test: Oral Health Habits — Tooth brushing frequency Dental floss usage Annual dentist visits
Diagnostic Test: Oral Findings — DMFT/dft Index: Measures decayed, missing, and filled teeth. ICDAS II: International Caries Detection and Assessment System, used for detecting and assessing dental caries.
  DDE Index: Developmental Defects of Enamel index. BAKH Index: Basic Anatomic Keratinization Hierarchy, typically used in specific studies.
  DI (Debris Index): Assesses oral hygiene based on the amount of debris on the teeth.
  CI (Calculus Index): Measures the amount of calculus (tartar) on the teeth. OHI-S (Simplified Oral Hygiene Index): Assesses oral hygiene based on the presence of debris and calculus.
  MGI (Modified Gingival Index): Assesses the severity of gingivitis based on inflammation.
Diagnostic Test: Quality of Life Assessment — KINDLR Scale: Used to assess disease-related quality of life from both the child's and the parent's perspectives.

SUMMARY:
The aim of this study is to compare the oral health findings, salivary parameters and disease-related quality of life of children with different stages of Chronic Kidney Disease(CKD), those undergoing dialysis and transplantation, with healthy children, and to evaluate certain serum biomarkers in children with CKD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a progressive and irreversible decline in the function of many nephrons and glomerular filtration rate due to kidney diseases. This decline leads to increased serum levels of urea and creatinine. Patients with CKD often exhibit various oral manifestations, such as an ammonia-like odor, gingival enlargement due to drug therapy, enamel hypoplasia, dental calculus, dry mouth, uremic stomatitis, and oral mucosal lesions. Interestingly, children with CKD tend to have a lower prevalence of dental caries, likely due to the high urea content in their saliva, which has antibacterial properties. CKD is also associated with salivary gland dysfunction and increased oxidative damage. Furthermore, CKD patients have reduced bone quality, making them more susceptible to fractures. A study on the quality of life (QoL) in children with CKD and their parents reported significantly lower physical and social QoL scores in children undergoing hemodialysis compared to healthy controls. This study aims to comparatively evaluate and analyze children diagnosed with different stages of chronic kidney disease (CKD) and healthy children without any systemic conditions, focusing on their age, gender, and oral health habits such as tooth brushing frequency, dental floss usage, and annual dentist visits. Disease-related information such as the stage of CKD, dialysis, and transplantation, as well as oral findings, will be examined using DMFT/dft, ICDAS II, DDE, BAKH, DI, CI, OHI-S, and MGI indices. The study will assess general disease-related quality of life from both the child's and the parent's perspectives using the KINDLR scale. Additionally, salivary samples collected from children with CKD and healthy children will be analyzed for salivary flow rate, pH, buffering capacity, total oxidant and antioxidant capacities, urea, calcium, potassium, and phosphorus levels. Serum urea, calcium, and phosphorus values will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Not having any systemic disease.
* Not being on any regular medication.

Exclusion Criteria:

* Having any systemic disease.
* Being on any regular medication.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Being followed up for a diagnosis of chronic kidney disease
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Oral Health Status | baseline
  DMFT/dft indices, DI (Debris Index), CI (Calculus Index), and OHI-S (Simplified Oral Hygiene Index) scores,DDE Index (Developmental Defect of Enamel), MGI Index (Modified Gingival Index) and ICDAS-II. DMFT/dft index values, DI, CI, and OHI-S scores as numerical values. DDE, MGI Index and ICDAS-II are percentage of participants with these conditions. Prevalence of limited opacities, caries and gingival inflammation based on DDE, ICDAS II and MGI indices.
Salivary Analysis | baseline
  Salivary urea, calcium (Ca), potassium (K), phosphorus (P), total oxidant status (TOS) levels, and salivary flow rate. Concentration of urea, Ca, K, P, TOS in mg/dL or equivalent, and salivary flow rate in mL/min.
Quality of Life (QoL) | baseline
  Quality of life scores on the KINDLR scale for both children with CKD and their parents

SECONDARY OUTCOMES:
Correlation Between Oral Health Indices and Salivary Biomarkers | baseline
  Correlation between DMFT/dft index, DI, CI, OHI-S scores, and salivary levels of urea, calcium (Ca), potassium (K), phosphorus (P), total oxidant status (TOS), and total antioxidant status (TAS). Pearson or Spearman correlation coefficient. DMFT/dft index, DI, CI, OHI-S scores for oral health assessment; biochemical analysis for salivary biomarker levels.
Correlation Between Salivary Urea and Serum Urea Levels | baseline
  Correlation between salivary urea levels and serum urea levels. Pearson or Spearman correlation coefficient. Biochemical analysis for salivary and serum urea levels.
Correlation Between Salivary and Serum Calcium and Phosphorus Levels: | baseline
  Correlation between salivary calcium and phosphorus levels and serum calcium and phosphorus levels. Pearson or Spearman correlation coefficient. Biochemical analysis for salivary and serum calcium and phosphorus levels.

CONTACTS AND LOCATIONS:
Overall Officials: Harika Alpay, Prof, Study Chair — Marmara University Faculty of Medicine; İbrahim Gökçe, Prof, Study Chair — Marmara University Faculty of Medicine; Nurdan Yıldız, Prof, Study Chair — Marmara University Faculty of Medicine; Nihal Şehkar Oktay, Assoc. Prof, Study Chair — Marmara University Faculty of Medicine
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Maltepe, Turkey (Türkiye)

REFERENCES:
- [Derived] Kodaman Dokumacigil N, Sezer B, Oktay S, Alpay H, Kargul B. Dental caries, oral hygiene and salivary characteristics in children with chronic kidney disease: a case-control study. Pediatr Nephrol. 2025 Aug;40(8):2627-2637. doi: 10.1007/s00467-025-06730-4. Epub 2025 Mar 19. PMID 40105933